CLINICAL TRIAL: NCT06351150
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase III Trial to Evaluate the Efficacy and Safety of Angiotensin II Injection in the Background Treatment of Catecholamines and Other Vasopressors in Chinese Adult Patients With Refractory Distributive Shock
Brief Title: Efficacy and Safety of Angiotensin II Injection Versus Placebo in Patients With Refractory Distributed Shock
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQG3902-III-01
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-04

CONDITIONS: Vasodilatory Shock
MeSH Terms: interventions — Angiotensin II; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angiotensin Ⅱ Injection (Experimental): Angiotensin II injection is administered via central vein, and the drug dosage is adjusted according to Mean Arterial Pressure (MAP), with an allowable dose of 1.25~160 ng/kg/min. Maximum 168 h.
  Interventions: Drug: Angiotensin II Injection
- Placebo (Placebo Comparator): The placebo is administered via central vein, and the drug dosage is adjusted according to MAP, with an allowable dose of 1.25~160 ng/kg/min. Maximum 168 h.
  Interventions: Drug: 0.9% sodium chloride injection

INTERVENTIONS:
Drug: Angiotensin II Injection — 1、Angiotensin II injection is a naturally occurring octapeptide hormone in the human renin angiotensin aldosterone system (RAAS). It is the main effector molecule of the RAAS system and one of the strongest known vasoconstrictors, involved in neurohumoral regulation.
  Arms: Angiotensin Ⅱ Injection
Drug: 0.9% sodium chloride injection — 0.9% sodium chloride injection, not containing active ingredients.
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled study on the treatment of refractory distributed shock with angiotensin II injection, with a random ratio of 1:1. Assuming a success rate of 25% for the main therapeutic endpoint in the control group and 50% for the experimental group, a total of 214 subjects will be enrolled, including 107 in the experimental group and 107 in the control group.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 years to 75 years old, male or female;
* diagnosis of distributive shock;
* on the basis of the treatment of total vasoactive drugs dose > 0.2 μg/kg/min norepinephrine (or equivalent dose of another vasoactive drug: such as epinephrine > 0.2 μg/kg/min, dopamine > 30 μg/kg/min, phenylephrine > 2 μg/kg/min, vasopressin > 0.08 U/min) and continuous treatment for at least 6 hours and no more than 48 hours, the patient's mean arterial pressure can still only be maintained between 55 and 70 mmHg, or do not reach the target MAP assessed by clinicians, it can be diagnosed as refractory distributive shock.
* have central venous access and arterial catheters, and are expected to be present for at least the first 48 hours of the study.
* indwelling catheter, and expected to be present for at least the first 48 hours of the study.
* patient has received at least 30 mL/kg of crystalloid or colloid volume in the previous 24 hours or has undergone adequate volume resuscitation in the opinion of the investigator.
* patients must have one of the following criteria with clinical features of high-output shock

  1. Central venous oxygen saturation (ScVO2) > 70% (via saturation catheter or central venous blood gas) and central venous pressure (CVP) > 8 mmHg.
  2. cardiac index (CI) > 2.3 L/min/m2.
* the patient or legal representative is willing and able to provide written informed consent and comply with all protocol requirements.

Exclusion Criteria:

* Patients with burns > 20% of total body surface area;
* Patients with cardiovascular (CV) SOFA score ≤ 3;
* Patients with acute coronary syndrome requiring interventional therapy;
* Patients treated with Extracorporeal Membrane Oxygenation (ECMO);
* Patients with end-stage liver failure (Model for end-stage liver disease score (MELD) > 30).
* Patients with a diagnosis of asthma or bronchospasm.
* Patients with a diagnosis of acute mesenteric ischemia, or patients with suspected acute mesenteric ischemia.
* Patients with a history, presence, or high suspicion of aortic dissection or abdominal aortic aneurysm, or patients diagnosed with aortic dissection or abdominal aortic aneurysm.
* Patients who have been diagnosed with malignant tumor within the past 2 years, except for early malignant tumors (carcinoma in situ or stage I tumor) that have been radically treated or expected to recover after treatment, such as adequately treated thyroid cancer, cervical carcinoma in situ, basal cell or squamous cell carcinoma.
* Patients with Raynaud's phenomenon, systemic sclerosis or vasospastic disease.
* Patients with life expectancy ≤ 24 hours as assessed by the study physician.
* Patients with active bleeding who are expected to require transfusion of > 4 units of packed red blood cells within 48 hours of study start.
* Patients with active bleeding and hemoglobin < 7 g/dL or any other condition that contraindicates serial blood sampling.
* Patients with absolute neutrophil count (ANC) < 1000 cells/mm3.
* Patients with known hypersensitivity to angiotensin II injection and its excipients.
* Patients who are currently participating in another interventional clinical trial.
* Blood/urine pregnancy test should be performed for patients with known pregnancy at screening and those with clinical suspicion of pregnancy.
* Patients who are considered unstable by the investigator or have any condition that would affect the safety of the study or the interpretation of the study results, or that would prevent the patient from completing the study, including but not limited to cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical disorders. For example: patients with arrhythmia, uncontrolled hyperglycemia, cerebrovascular disease, uncontrolled hypertension, autoimmune disease requiring daily use of ≥ 500 mg hydrocortisone or equivalent glucocorticoids, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with blood pressure response at 3 hours after administration of study drug | 3 hours after dose
  Defined as MAP ≥ 75 mmHg or MAP increase ≥ 10 mmHg from baseline compared to baseline without an increase in the dose of background vasoactive agents

SECONDARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) total score | 48 hours after dose
  Change from baseline in Sequential Organ Failure Assessment (SOFA) total score. The SOFA score evaluates organ failure according to the conditions of respiratory, blood, liver, cardiovascular, central nervous, kidney and other systems, is scored from 0 to 4, with a higher score representing more severe failure.
Cardiovascular SOFA subscore | 48 hours after dose
  Change from baseline in Sequential Organ Failure Assessment (SOFA) subscore. The SOFA score evaluates organ failure according to the conditions of respiratory, blood, liver, cardiovascular, central nervous, kidney and other systems, is scored from 0 to 4, with a higher score representing more severe failure.
Mortality at Day 7 | Day 7 after dose
  All-cause mortality of subject at Day 7
Mortality at Day 28 | Day 28 after dose
  All-cause mortality of subject at Day 28
Proportion of subjects with blood pressure response at 1 hour after administration | 1 hour after dose
  Defined as MAP ≥ 75 mmHg or MAP increase ≥ 10 mmHg from baseline compared to baseline without an increase in the dose of background vasoactive agents
Proportion of subjects with blood pressure response at 2 hours after administration | 2 hours after dose
  Defined as MAP ≥ 75 mmHg or MAP increase ≥ 10 mmHg from baseline compared to baseline without an increase in the dose of background vasoactive agents
Change in background vasoactive agent dose from 0 to 48 hours | 48 hours after dose
  Change in background vasoactive dose from baseline to 48 hours after dose
Absolute change in blood lactate from 0 to 3 hours | 3 hours after dose
  Absolute change in blood lactate from 0 to 3 hours
Absolute change in blood lactate from 3 to 48 hours | 3 to 48 hours after dose
  Absolute change in blood lactate from 3 to 48 hours
Absolute change in heart rate from 0 to 3 hours | 3 hours after dose
  Absolute change in heart rate from 0 to 3 hours
Absolute change in heart rate from 3 to 48 hours | 3 to 48 hours after dose
  Absolute change in heart rate from 3 to 48 hours
Adverse events (AE) | From drug administration to the end of the study, a total of 28 days
  Incidence and severity of adverse events (AE)
Serious adverse events (SAE) | From drug administration to the end of the study, a total of 28 days
  Incidence and severity of serious adverse events (SAE)

CONTACTS AND LOCATIONS:
Locations (42):
- China (42):
  - The Second People's Hospital of Hefei, Hefei, Anhui
  - The Frist Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Tiantan Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The Frist Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The people's Hospital of the University of traditional Chinese medicine in Fujian, Fuzhou, Fujian
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Sun Yat sen University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Qingyuan Hospital Affiliated to Guangzhou Medical University, Qingyuan, Guangdong
  - The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Guilin, Guangxi
  - Liuzhou General Hospital, Liuchow, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Affiliated Hospital of Hebei University, Baoding, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College of huazhong university of science and technology, Wuhan, Hubei
  - Wuhan Third Hospital, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The Frist Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Frist Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Frist Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - Taizhou hospital of Zhejiang Province, Taizhou, Zhejiang